CLINICAL TRIAL: NCT03493269
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess Safety, Tolerability, Pharmacokinetics and Exploratory Pharmacodynamics of Multiple Oral Doses of BAY1834845 in Healthy Male Subjects and in Female and Male Patients With Psoriasis Over an Extended Treatment Duration
Brief Title: A Multiple Dose Study of BAY1834845 in Healthy Male Subjects and in Patients With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18385; 2017-001817-10 (EudraCT Number)
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — zabedosertib; Midazolam

STUDY DESIGN:
Intervention Model Description: Double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BAY1834845 (Experimental): Part 1 in healthy male subjects:
  Dose Groups 1-4 : orally administered multiple ascending doses. The treatment will last 10 consecutive days (treatment period1) and 1 day (treatment period 2) Dose Group 5: The treatment will last 1 day (treatment period 1) and 10 consecutive days (treatment period 2)
  Interventions: Drug: BAY1834845; Drug: Midazolam
- Matching Placebo (Placebo Comparator): Part 1: Matching placebo in healthy male subjects.
  Interventions: Other: Matching Placebo; Drug: Midazolam
- Chosen dose of BAY1834845 (Experimental): Part 2: This dose level will be adminstered in female and male patients with psoriasis
  Interventions: Drug: BAY1834845
- Placebo (Placebo Comparator): Part 2: The placebo will be adminstered in female and male patients with psoriasis
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: BAY1834845 — Orally administered.
  Arms: BAY1834845; Chosen dose of BAY1834845
Other: Matching Placebo — Orally administered.
  Arms: Matching Placebo; Placebo
Drug: Midazolam — Part 1: Orally administered 1mg as a single dose.
  Arms: BAY1834845; Matching Placebo

SUMMARY:
To assess safety and tolerability of multiple oral doses of BAY1834845 in healthy male subjects (Part 1) and in patients with psoriasis (Part 2).

To assess the pharmacokinetic (PK) properties of total BAY1834845 in plasma after oral multiple doses of BAY1834845 in healthy male subjects (Part 1) and patients with psoriasis (Part 2).

ELIGIBILITY:
Inclusion Criteria:

Part 1 (healthy male subjects)

* Healthy male subjects, 18 to 50 years of age (inclusive), and in good health as determined by medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory tests at screening
* Body mass index (BMI) above or equal to 18.5 and lower or equal to 30 kg/m2 (BMI = body weight (kg) / [height (m)]2 and a body weight above or equal 50 kg Part 2 (patients with psoriasis)
* Male patients, 18 to 70 years of age (inclusive) or female patients of non-child bearing potential, 30 to 70 years of age (inclusive)
* Body mass index above or equal to 18.5 and lower or equal to 35 kg/m*2 and a body weight above 50 kg
* A documented diagnosis of psoriasis, with a history of at least 6 months prior to study drug administration. Moderate to severe plaque psoriasis at screening, defined by: a) an involved body surface area (BSA) above or equal to 10% of BSA, b) a Psoriasis Area and Severity Index (PASI) score of above or equal, 12 c) a Physician's Global Assessment (PGA) score of above or equal 2.

Exclusion Criteria:

* History of hypersensitivity to any of the components of the study drug
* Any clinically relevant abnormal findings in safety laboratory parameters and ECG
* History of tuberculosis (TB) or active or latent tuberculosis
* Receipt of live or attenuated vaccine 90 days prior to the first dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAEs) | Approximately 47 days
  Part 1 in healthy male subject
Severity of treatment-emergent adverse events (TEAEs) | Approximately 47 days
  Part 1 in healthy male subject
Frequency of treatment-emergent adverse events (TEAEs) | Approximately 84 days
  Part 2: Patients with psoriasis
Severity of treatment-emergent adverse events (TEAEs) | Approximately 84 days
  Part 2: Patients with psoriasis
AUC(0-24)md of BAY1834845 | Part 1 - Period 1 (dose group 1-4): Day 1 to 2 Part 1 - Period 2 (dose group 5): Day 1 to 2
  Part 1 AUC(0-24)md: AUC from zero to 24 hours after multiple dosing
AUC(0-12)md of BAY1834845 | Part 1 - Period 1 (dose group 1-4): Day 1, Part 1 - Period 2 (dose group 5): Day 1
  Part 1 AUC(0-12)md:AUC from zero to 12 hours after multiple dosing
Cmax,md of BAY1834845 | Part 1 - Period 1 (dose group 1-4): Day 1, Part 1 - Period 2 (dose group 5): Day 1
  Part 1 Cmax,md:Cmax(Maximum observed drug concentration, directly taken from analytical data) after multiple dosing
Cav,md of BAY1834845 | Part 1 - Period 1 (dose group 1-4): Day 1 to 2 Part 1 - Period 2 (dose group 5): Day 1 to 2
  Part 1 Cav:Average concentration within a dosing interval after multiple dosing
AUC(0-24)md of BAY1834845 | Part 2: one day between day 35 and 42
  Part 2: AUC(0-24)md: AUC from zero to 24 hours after multiple dosing
AUC(0-12)md of BAY1834845 | Part 2: one day between day 35 and 42
  Part 2: AUC(0-12)md: AUC from zero to 12 hours after multiple dosing
Cmax,md of BAY1834845 | Part 2: one day between day 35 and 42
  Part 2: Cmax,md:Cmax (Maximum observed drug concentration, directly taken from analytical data) after multiple dosing
Cav, md of BAY1834845 | Part 2: one day between day 35 and 42
  Part 2: Cav: Average concentration within a dosing interval after multiple dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Charité Research Organisation GmbH, Berlin
  - PAREXEL GmbH, Berlin

REFERENCES:
- [Derived] Feldmuller M, Jodl SJ, Ploeger B, Wagenfeld A, Wiesinger H, Zollmann FS, Klein S, Zhang R, Rohde B, Hochel J. Zabedosertib, a novel interleukin-1 receptor-associated kinase-4 inhibitor, shows a favorable pharmacokinetic and safety profile across multiple phase 1 studies. Front Pharmacol. 2025 May 30;16:1521505. doi: 10.3389/fphar.2025.1521505. eCollection 2025. PMID 40520205